CLINICAL TRIAL: NCT06289452
Title: An Open-label, Dose-escalation Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of IVB102 Injection in Subjects With X-linked Retinoschisis (XLRS)
Brief Title: Safety and Efficacy Study of IVB102 Injection in Subjects With X-linked Retinoschisis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: InnoVec Biotherapeutics Inc. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IVB102-101
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Retinoschisis; Retinal Disease; Retinal Degeneration; Eye Diseases
MeSH Terms: conditions — Retinoschisis; Retinal Diseases; Retinal Degeneration; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IVB102 Treatment Arm（Low dose） (Experimental): Intraocular injection of a single low dose of IVB102
  Interventions: Genetic: IVB102 Injection
- IVB102 Treatment Arm（Intermediate dose） (Experimental): Intraocular injection of a single intermediate dose of IVB102
  Interventions: Genetic: IVB102 Injection
- IVB102 Treatment Arm（High dose） (Experimental): Intraocular injection of a single high dose of IVB102
  Interventions: Genetic: IVB102 Injection

INTERVENTIONS:
Genetic: IVB102 Injection — Gene transfer by intravitreal injection of the RS1 AAV vector
  Arms: IVB102 Treatment Arm（Low dose）
Genetic: IVB102 Injection — Gene transfer by intravitreal injection of the RS1 AAV vector
  Arms: IVB102 Treatment Arm（Intermediate dose）
Genetic: IVB102 Injection — Gene transfer by intravitreal injection of the RS1 AAV vector
  Arms: IVB102 Treatment Arm（High dose）

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of IVB102 injection in subjects with XLRS.

DETAILED DESCRIPTION:
This is a open label, dose escalation, single-center study. One eye of each participant will receive a single IVB102 injection by intravitreal injection. Participants will be followed for 52 weeks after which they will continue to be followed for up to 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing and able to provide written, signed informed consent.
2. Male individual at least 8 years of age with clinical diagnosis of XLRS caused by mutations in RS1.
3. Best corrected visual acuity (BCVA) in the study eye of less than or equal to 63 (corresponding to a Snellen acuity of 20/63).
4. Must agree to use effective barrier (male or female condom) of contraception before dosing and continuing one year after gene transfer.

Exclusion Criteria:

1. Lens, cornea, or other media opacities in the study eye that preclude adequate visualization and testing of the retina.
2. Pre-existing eye conditions that would contribute significantly to visual loss or increase the risk of an intravitreal injection (e.g. DR、RVO or large retinal detachment).
3. Any intraocular surgery in the study eye within 6 months prior to screening.
4. Use of topical carbonic anhydrase inhibitors within 3 months prior to screening.
5. Use of anticoagulants or anti-platelet agents within 7 days prior to study agent administration.
6. Prior receipt of any AAV gene therapy product.
7. Use of any investigational agent within 3 months prior to screening.

Min Age: 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | 4 weeks
  Number and proportion of dose limited toxicity（DLTs）
Incidence of AEs | 52 weeks
  Number and severity of overall and ocular Adverse Events (AEs)
Incidence of SAEs | 52 weeks
  Number and severity of overall and ocular Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Visual function | 52 weeks
  Change from baseline in BCVA(Best Corrected Visual Acuity)(ETDRS)
OCT imaging | 52 weeks
  Change from baseline in CST(Central Retinal Thickness)(OCT)
ERG parameters | 52 weeks
  Change from baseline in response amplitudes measured using Electroretinogram (ERG)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pimenides D, George ND, Yates JR, Bradshaw K, Roberts SA, Moore AT, Trump D. X-linked retinoschisis: clinical phenotype and RS1 genotype in 86 UK patients. J Med Genet. 2005 Jun;42(6):e35. doi: 10.1136/jmg.2004.029769. PMID 15937075
- [Background] Wang XF, Chen FF, Zhou X, Cheng XX, Xie ZG. A novel mutation in RS1 and clinical manifestations in a Chinese twin family with congenital retinoschisis. Front Genet. 2022 Sep 23;13:993157. doi: 10.3389/fgene.2022.993157. eCollection 2022. PMID 36212125
- [Background] Sikkink SK, Biswas S, Parry NR, Stanga PE, Trump D. X-linked retinoschisis: an update. J Med Genet. 2007 Apr;44(4):225-32. doi: 10.1136/jmg.2006.047340. Epub 2006 Dec 15. PMID 17172462